CLINICAL TRIAL: NCT04986657
Title: A Prospective Study of Whole Genome Sequencing (ChromoSeq) as an Adjunct to Conventional Genomic Profiling in AML and MDS
Brief Title: Whole Genome Sequencing (ChromoSeq) as an Adjunct to Conventional Genomic Profiling in AML and MDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202105123
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Whole Genome Sequencing; Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Patients: ChromoSeq (Experimental): ChromoSeq will be performed on bone marrow DNA from consented patients in parallel with the standard of care cytogenetics, FISH, and the MyeloSeq gene panel obtained from that sample, in a CLIA licensed environment using CLIA-compliant ChromoSeq procedures.
  Interventions: Device: ChromoSeq
- Stakeholders (Treating Physicians) (No Intervention): -Stakeholders (treating physicians) will complete surveys/questionnaires. As of protocol amendment 10/31/2023, the stakeholders (treating physicians) will no longer be completing surveys/questionnaires.

INTERVENTIONS:
Device: ChromoSeq — Novel, streamlined whole genome sequencing approach
  Arms: Patients: ChromoSeq

SUMMARY:
This is a single institution, prospective study of the whole genome sequencing assay, ChromoSeq. Using prospectively collected patient data, coupled with physician surveys, the investigators seek to determine the feasibility of implementing ChromoSeq in addition to standard genomic testing, for patients with the diagnoses of acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria Patient

* Patient with a clinical suspicion for a new diagnosis of AML or MDS for whom the diagnostic molecular testing via the hematologic molecular algorithm (HMA) at BJH is requested or planned to be requested.
* Adult patients 18 years or older.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Inclusion Criteria Physician

* Treating physician at Washington University School of Medicine who directs therapy for individuals with hematologic malignancies.
* Able and willing to complete standardized questionnaires about usability, and stakeholder perceptions of ChromoSeq during the ChromoSeq implementation process.

Exclusion Criteria Patient

* Younger than 18 years of age

Exclusion Criteria Physician

* Does not treat patients at Washington University School of Medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of ChromoSeq as measured by total number of recurrent structural variants identified | Through completion of all ChromoSeq tests (estimated to be 15 months)
  * As compared to conventional cytogenetics in a real-time clinical setting
  * The total number of recurrent structural variants will be measured in each sample by ChromoSeq and metaphase cytogenetics yielding a pair of measurements. Each measurement will also be dichotomized into the presence or absence of at least one recurrent structural variant. The hypothesis of no difference in the number of variants detected by each method will be analyzed by a paired-sample t-test. However, if it is determined that the assumptions of a t-test are not tenable then a paired-sample sign test will be used instead. McNemar's test will be used to compare whether or not at least one recurrent structural variant identified is by each method.
Sensitivity of ChromoSeq as measured by total number of copy number alterations identified | Through completion of all ChromoSeq tests (estimated to be 15 months)
  * As compared to conventional cytogenetics in a real-time clinical setting
  * The total number of copy number alterations will be measured in each sample by ChromoSeq and metaphase cytogenetics yielding a pair of measurements. Each measurement will also be dichotomized into the presence or absence of at least one copy number alteration. The hypothesis of no difference in the number of copy number alterations detected by each method will be analyzed by a paired-sample t-test. However, if it is determined that the assumptions of a t-test are not tenable then a paired-sample sign test will be used instead. McNemar's test will be used to compare whether or not at least one copy number alterations is identified is by each method.
Sensitivity of ChromoSeq as measured by number of single nucleotide variants identified | Through completion of all ChromoSeq tests (estimated to be 15 months)
  * As compared to high coverage gene panels in a real-time clinical setting
  * The number of single nucleotide variants will be counted for each sample. Additionally, the data will be dichotomized into the presence or absence of at least one single nucleotide variant. Data will be analyzed by paired-sample t-tests and McNemar's test.
Sensitivity of ChromoSeq as measured by number of insertion-deletions identified | Through completion of all ChromoSeq tests (estimated to be 15 months)
  * As compared to high coverage gene panels in a real-time clinical setting
  * The number of insertion-deletions will be counted for each sample. Additionally, the data will be dichotomized into the presence or absence of at least one insertion-deletion. Data will be analyzed by paired-sample t-tests and McNemar's test.
Determine if risk-stratification using ChromoSeq correlates with overall-survival | Through completion of follow-up for all patients (estimated to be 63 months)
  * As compared to metaphase cytogenetics
  * The relationship of risk-stratification defined by either ChromoSeq or conventional cytogenetics to clinical outcome will be illustrated with Kaplan-Meier survival analyses on overall survival for both ChromoSeq and metaphase cytogenetics. The predictive accuracy of the two methods will be tested by comparing the area under the ROC curves using the method of DeLong et al.
Determine if risk-stratification using ChromoSeq correlates with event-free survival | Through completion of follow-up for all patients (estimated to be 63 months)
  * As compared to metaphase cytogenetics
  * The relationship of risk-stratification defined by either ChromoSeq or conventional cytogenetics to clinical outcome will be illustrated with Kaplan-Meier survival analyses on event-free survival for both ChromoSeq and metaphase cytogenetics. The predictive accuracy of the two methods will be tested by comparing the area under the ROC curves using the method of DeLong et al.
Proportion of cases in which ChromoSeq provides new genetic information to the clinician | Through completion of all ChromoSeq tests (estimated to be 15 months)
  * As compared to conventional genomic profiling (cytogenetics, FISH, and next-generation sequencing) that is used for clinical management (such as risk-stratification or institution of targeted gene therapy)
  * Items in the ChromoSeq Implementation Physician Survey will be used to describe physician evaluation of ChromoSeq with conventional genomic profiling with regard to clinical management. Responses to these items will be presented in frequency tables. For statistical analysis, the values of each item will be recoded from 1-5 to -2 to +2 and one-sample t-tests used to test the null hypothesis that the mean value is 0 (neither agree nor disagree.) In addition, case-reports will be reviewed for qualitative evaluations of physician experience with the two methods.
ChromoSeq turnaround time | Through completion of all ChromoSeq tests (estimated to be 15 months)
  -Measured from time of order requisition (hematologic molecular algorithm from Barnes Jewish Hospital) to return of report to the medical record
Proportion of failed ChromoSeq assays | Through completion of all ChromoSeq tests (estimated to be 15 months)
  * As compared to failed standard of care genomic profiling assays
  * Each assay will be categorized as successful or failed and a two-way table constructed displaying ChromoSeq assay status by standard assay status. A Pearson chi-square test will be calculated to test the null hypothesis that assay success is independent of type of assay.

SECONDARY OUTCOMES:
Stakeholder perceptions of ChromoSeq | Within 1 month after generation of ChromoSeq (estimated to be 2 months)
  * Using survey responses from treating physicians obtained from per case standardized questionnaires designed using Consolidated Framework for Implementation Research constructs
  * For each case, the corresponding treating physician will be asked to answer a case-based ChromoSeq Implementation Physician Survey. In order to prospectively investigate how the ChromoSeq data was used or could be used by the treating physician for each case, and to evaluate perceptions in real time, the physician will be asked to complete the survey within 1 month of the ChromoSeq and completed conventional genomic profiling results being returned to the chart, whichever is later.
Stakeholder perceptions of ChromoSeq as measured by the Acceptability of Intervention Measure | When 100 genomes have been sequenced (estimated to be 12 months)
  * Will complete survey at the time when 100 genomes have been sequenced
  * 4 statements with answers ranging from 1=completely disagree to 5=completely agree.
Stakeholder perceptions of ChromoSeq as measured by the Intervention Appropriateness Measure | When 100 genomes have been sequenced (estimated to be 12 months)
  * Will complete survey at the time when 100 genomes have been sequenced.
  * 4 statements with answers ranging from 1=completely disagree to 5=completely agree.
Stakeholder perceptions of ChromoSeq as measured by the Feasibility of Implementation Measure | When 100 genomes have been sequenced (estimated to be 12 months)
  -Will complete survey at the time when 100 genomes have been sequenced.
  --4 statements with answers ranging from 1=completely disagree to 5=completely agree.
Stakeholder perceptions of ChromoSeq as measured by the System Usability Scale | When 100 genomes have been sequenced (estimated to be 12 months)
  * Will complete survey at the time when 100 genomes have been sequenced.
  * 10 statements about usability of ChromoSeq with answers ranging from 1=strongly disagree to 5=strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Meagan Jacoby, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal may submit proposals to mjacoby@wustl.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu